CLINICAL TRIAL: NCT00213785
Title: A Study of Plasmatic Concentrations of Endothelin-1 (ET1), Atrial Natriuretic Peptide (ANP) and Brain Natriuretic Peptide (BNP) in Acute Ischemic Stroke.
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Other Study IDs: 2558
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Stroke
Keywords: AreET1; ANP; BNP pronostic markers of stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
A study of plasmatic concentrations of endothelin-1 (ET1), atrial natriuretic peptide (ANP) and brain natriuretic peptide (BNP) in acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age > 18
* with an ischemic stroke

Exclusion Criteria:

* cardiac failure
* renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2001-11; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Andoni Echanz-Laguna, MD, Principal Investigator — Hopitaux Universitaires de Strasbourg
Locations (1):
- Clinique neurologique - Service des maladies du système nerveux et du muscle - Hôpitaux Universitaires de Strasbourg, Hôpital Civil, Strasbourg, France